CLINICAL TRIAL: NCT04099277
Title: A Phase 1a/1b Study of LY3435151 Administered to Patients With Advanced Solid Tumors
Brief Title: A Study of LY3435151 in Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to strategic business decision by Eli Lilly and Company.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17364; J1Q-MC-JZIA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor; Triple-negative Breast Cancer; Gastric Adenocarcinoma; Head and Neck Squamous Cell Carcinoma; Cervical Carcinoma; High Grade Serous Ovarian Carcinoma; Hepatocellular Carcinoma; Undifferentiated Pleomorphic Sarcoma; Leiomyosarcoma
Keywords: immunotherapy; CD226 agonist
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Histiocytoma, Malignant Fibrous; Leiomyosarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: 10 milligrams (mg) LY3435151 (Experimental): Participants received intravenous (IV) push or IV bolus infusion of 10 mg LY3435151.
  Interventions: Drug: LY3435151
- Part B: LY3435151 + Pembrolizumab Dose Escalation (Experimental): Pembrolizumab was not administered as study was terminated before completion of Part A of the dose escalation period.
  Interventions: Drug: LY3435151; Drug: Pembrolizumab
- Part C: LY3435151 Dose Expansion (Experimental): Participants were not enrolled in to this arm, as trial was terminated in dose escalation phase.
  Interventions: Drug: LY3435151
- Part D: LY3435151 + Pembrolizumab Dose Expansion (Experimental): Participants were not enrolled in to this arm, as trial was terminated in dose escalation phase.
  Interventions: Drug: LY3435151; Drug: Pembrolizumab

INTERVENTIONS:
Drug: LY3435151 — Administered IV
Drug: Pembrolizumab — Administered IV
  Arms: Part B: LY3435151 + Pembrolizumab Dose Escalation; Part D: LY3435151 + Pembrolizumab Dose Expansion

SUMMARY:
The reason for this study is to see if the study drug LY3435151 is safe in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have certain types of cancer, which your study doctor will discuss with you
* Participant must have stopped other forms of treatment for cancer, which your study doctor will discuss with you
* Participant must be able and willing to provide a sample of your tumor before beginning treatment and once while on treatment. For certain tumor types, the outcome of the biopsy may exclude you from the study treatment (for Phase 1b)
* Participant must agree to use birth control
* Participant must have progressed through or are intolerant to therapies with known clinical benefit, which your study doctor will discuss with you

Exclusion Criteria:

* Participant must not have a history of tuberculosis, uncontrolled HIV or uncontrolled hepatitis B or C virus infection
* Participant must not have an autoimmune disease, which your study doctor will discuss with you
* Participant must not use corticosteroids, which your study doctor will discuss with you
* Participant must not have heart disease, Crohn's disease or brain cancer
* Participant must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- National Cancer Center Hospital, Chuo-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3435151 in Participants With Solid Tumors — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JZIA#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg LY3435151: Participants received 10 milligrams (mg) dose of LY3435151 via intravenous (IV) as an IV push or IV bolus infusion.
Period: Overall Study
Arm/Group | 10 mg LY3435151
Started | 2
Received at Least 1 Dose of Study Drug | 2
Completed | 0
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 10 mg LY3435151: Participants received 10 mg dose of LY3435151 via intravenous (IV) as an IV push or IV bolus infusion.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1
  Japan | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With LY3435151 Dose-Limiting Toxicities (DLTs)
Description: A DLT is defined as an Adverse Event that is likely related to the study medication or combination, and fulfills any one of the following criteria, graded according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0:
  1. Any death not clearly due to the underlying disease or extraneous causes
  2. Neutropenic fever 2. Any Grade ≥3 non-hematologic toxicity
  3. Grade ≥4 neutropenia or thrombocytopenia >7 days
  4. Grade ≥3 thrombocytopenia with bleeding
  5. Grade ≥3 nausea/vomiting or diarrhea>72 hours with adequate antiemetic and other supportive care
  6. Grade ≥3 fatigue ≥1 week
  7. Grade ≥3 electrolyte abnormality that lasts>72 hours, unless the Participant has clinical symptoms, in which case all Grade 3+electrolyte abnormality regardless of duration should count as a DLT
  8. Grade ≥3 prolongation of QT interval corrected using the Fridericia formula on 2 separate electrocardiogram readings approximately 5 min apart.
Time Frame: Baseline through Cycle 2 (21 Day Cycles)
Population: Zero participants were analyzed. This outcome was not determined because the study terminated before completion of Part A of the dose escalation period.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3435151
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3435151.
Time Frame: Cycle 1 Day 1 (C1D1) (Predose, 1, 3 hour (hr), C1D2 (24 hr), C1D4 (72hr), C1D8 (168hr), C1D15 (336hr)
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 2
microgram per milliliter (µg/mL) | NA (NA) — 2.07, 7.16 (Individual values reported as there were only two participants)

3. Secondary Outcome: PK: Cmax of LY3435151 in Combination With Pembrolizumab
Description: PK: Cmax of LY3435151 in Combination with Pembrolizumab.
Time Frame: Predose Cycle 1 Day 1 through Predose Cycle 5 Day 1 (21 Day Cycles)
Population: Zero participants were analyzed. The study was terminated early and no data was collected.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants With Complete Response (CR) or Partial Response (PR)
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the independent central review according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants per cohort with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline through Disease Progression or Death (Up to 4 Months)
Population: Zero participants were analyzed. The study was terminated early and no data was collected.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, and Stable Disease
Description: Disease Control Rate (DCR) is the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline through Measured Progressive Disease (Up to 4 Months)
Population: Zero participants were analyzed. The study was terminated early and no data was collected.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response (DoR)
Description: DOR is the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up to 4 Months)
Population: Zero participants were analyzed. The study was terminated early and no data was collected.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) is defined as the time from the date of start of treatment to the date measurement criteria for confirmed CR or PR (whichever is first recorded) are first met. For participants who are not known to have achieved CR or PR as of the data inclusion cut-off date, TTR will be censored at the date of the last objective disease assessment prior the date of any subsequent systematic anticancer therapy.
Time Frame: Baseline to Date of CR or PR (Up to 4 Months)
Population: Zero participants were analyzed. The study was terminated early and no data was collected.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS time was measured from the date of randomization until the first radiographic documentation of progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Baseline to Objective Progression or Death Due to Any Cause (Up to 4 Months)
Population: Zero participants were analyzed. The study was terminated early and no data was collected.
Arm/Group | 10 mg LY3435151
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 Months
Description: All randomized participants.
Arm/Group | 10 mg LY3435151
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg LY3435151 (N=2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg LY3435151 (N=2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1)
Troponin i increased (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated before completion of the dose escalation phase (Part A), due to strategic business decision made by the company.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT04099277/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT04099277/SAP_001.pdf